CLINICAL TRIAL: NCT01893710
Title: International (Pediatric) Peritoneal Biobank
Status: Recruiting | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Claus Peter Schmitt, MD, Heidelberg University
Other Study IDs: IPPB Biobank; University of Heidelberg (Other: University of Heidelberg, Medical Faculty)
Record Dates: First submitted 2013-06-27; First posted 2013-07-09 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Kidney Failure, Chronic; Peritoneal Dialysis Complication; Transplantation; Healthy
Keywords: peritoneal dialysis; parietal peritoneum; omentum; chronic kidney disease; vasculopathy
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Vascular Diseases | interventions — Chorionic Villi Sampling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Parietal ond omental peritoneal membrane specimen will be collected in all groups
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control: 'Biopsy sampling': Peritoneal biopsies without kidney disease, i.e. diseases not related to the kidney and not affecting the peritoneum. This group is accomplished.
- chronic kidney disease: Samples will obtained from patients with chronic kidney disease stage 5 (at time of catheter Insertion)
  Interventions: Procedure: biopsy sampling
- Peritoneal dialysis: Patients on PD with different PD fluids and intercurrent abdominal surgery and at time of renal transplantation.
  Interventions: Procedure: biopsy sampling
- Post PD and with functioning graft: Samples will also be collected and analysed from patients with renal transplantation after PD at time of and tenckhoff catheter removal several weeks after Tx or other intercurrent abdominal surgery.
  Interventions: Procedure: biopsy sampling

INTERVENTIONS:
Procedure: biopsy sampling — Two parietal peritoneal samples, each 1 cm² x 0.3 cm in depth and three omental tissue samples, each 1 cm² in size will be obtained.
  Biopsy sampling will be performed in all groups. This is an observational not an interventional trial.
  Groups: Peritoneal dialysis; Post PD and with functioning graft; chronic kidney disease

SUMMARY:
Within few years the peritoneal membrane of adult peritoneal dialysis (PD) patients undergoes substantial morphological transformation, including progressive fibrosis, vasculopathy and neoangiogenesis. Ultrafiltration capacity steadily declines and ultimately results in PD failure. In children, peritoneal biopsies demonstrating PD associated alterations have not yet been obtained. They, however, should be particularly informative, since secondary tissue and vascular pathology related to ageing or diabetes is absent.

An international, prospective peritoneal membrane biopsy study in children on PD will therefore be performed. Biopsies will be obtained at time of PD catheter insertion, on occasion of intercurrent abdominal surgery (e.g. hernia repair, catheter exchange) and at time of renal transplantation. Quantitative histomorphometry and tissue protein expression analyses will be correlated with time integrated PD treatment modalities and functional characteristics as well as inflammatory and cardiovascular comorbidity surrogate parameter. Blood will be obtained during clinical routine sampling. Biopsies will be obtained during clinically indicated operations, without substantially increasing operation time and associated surgical risks. The detailed histomorphometry of the PD membrane will give additional information, potentially impacting on the individual PD regime.

3/2018: The analyses of the pediatric PD biopsy demonstrated early and major transformation of the peritoneal membrane with neutral pH low GDP fluids, and significant vasculopathy already in children with CKD stage 5, further progressing with PD. The underlying mechanisms are partly understood, only. In view of these major findings and the numerous open questions, collection of biosamples will be continued in children and also in adult PD patients. The following questions will be addressed: Molecular counterparts of peritoneal semi-permeability, solute and water transport (beyond AQP1), pathomechanisms and molecular and functional impact of peritoneal transformation with low and high GDP fluids, and the respective pathomechanisms and molecular and functional impact of vascular disease in CKD and with different PD fluids. The impact of renal transplantation following PD will be assessed in a subgroup of patients with tenckhoff catheter removal several weeks after transplantation and a functioning graft.

DETAILED DESCRIPTION:
Please see study protocol and

http://www.pedpd.org

ELIGIBILITY:
Inclusion Criteria

* Age 0 to 90 years
* CKD 5D, peritoneal dialysis and
* Patients with normal renal function and elective abdominal surgery due to limited abdominal pathology (such as hernia repair, gallstones….)
* Patients post PD and post Tx
* Oral and written consent
* Ability to consent of the adult patient and of the parents and legal guardian of patients not yet of legal age, respectively

Exclusion Criteria:

* Abdominal adhesions, malformation and inflammation beyond PD induced changes
* Patients with disseminated tumour disease
* Patients with critical heart failure and other medical conditions, where the additional procedure may confer an increased increase risk
* Pregnancy
* Preterm babies (below 37 weeks of gestational age)
* Serum hemoglobin < 10 g/dl in newborns and < 8 g/dl in children and adults

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: See eligibility data
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-02; Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Peritoneal vasculopathy (lumen vessel ratio) | Two years (Mean PD treatment time)
  Digital quantification of degree of vasculopathy, i.e the lumen vessel ratio. Healthy children have a L/V ratio of about 0.7. lower values represent vasculopathy with lumen narrowing, 0 is complete obliteration of the vessel.
  This measurements will be accompanied by molecular analysis of pathomechanisms (including omics Technology)

SECONDARY OUTCOMES:
Number of vessels per peritoneal membrane area (per mm²) | at time of catheter insertion, intercurrent abdominal surgery and at time of renal transplantation
  Digital histomorphometry of small vessel density per mm² submesothelial section area analysed.

OTHER OUTCOMES:
Submesothelial thickness (µm) | 2 years (average PD duration)
  Digital imaging analysis of submesothelial thickness as a marker of peritoneal fibrosis (distance between mesothelium and adjacent muscle/adipos tissue)
Submesothelial lymphocyte, macrophage, MMT cell count | 2 years (mean PD duration)
  Quantification of peritoneal leucocyte Infiltration, i.e. number of CD45 positive lymphocytes and CD68 positive macrophages per mm² of submesothelial section area . The number of cells that underwent mesothelial-mesenchymal transition per mm² submesothelial section are quantified by immunohistochemical co-staining of mesothelial and fibroblast marker (cytokeratin and FSP1).
Peritoneal VEGF and pSMAD abundance | 2 years (mean PD duration)
  Key cytokines involved in peritoneal membrane transformation will be measured immunohistochemically. These are VEGF and TGF-beta induced p-SMAD (%positive area per section area analysed).

CONTACTS AND LOCATIONS:
Overall Officials: Claus P Schmitt, MD, Principal Investigator — University of Heidelberg, Center for Pediatric and Adolescent Medicine
Locations (26):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Mercy Hospital, Kansas City, Missouri
  - The Children´s Hospital of Philadelphia, Narberth, Pennsylvania
- Department of Pediatrics, Medical University Vienna, Vienna, Austria
- UZ Ghent, Ghent, Belgium
- University Children's Hospital, Prague, Czechia
- France (2):
  - Service de Néphrologie Pédiatrique, Hôpital Femme Mere Enfant, Lyon
  - University Children's Hospital, Strasbourg
- Germany (6):
  - Department of Medicine I (Nephrology), University of Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Children's Hospital, Berlin
  - University Children's Hospital, Cologne
  - University Children's Hospital, Essen
  - UKE, University Children´s Hospital, Hamburg
  - KfH Pediatric Kidney Center, Department of Pediatric Nephrology, University of Marburg, Marburg
- University Children's Hospital, Budapest, Hungary
- Italy (3):
  - University Children'Hospital, Genova
  - University Children's Hospital, Milan
  - Pediatric Nephrology, Dialysis and Transplant Unit, Padua
- University children's Hospital, Vilnius, Lithuania
- Paediatric CAPD unit, Kuala Lumpur Hospital, Kuala Lumpur, Malaysia
- Krakow, Jagiellonian University Medical College, Krakow, Poland
- Hospital Universitario Materno-Infantil Vall d' Hebron, Barcelona, Spain
- Karolinska University Hospital, Stockholm, Sweden
- Children's Hospital, Inselspital, Bern University Hospital and University of Bern, Bern, Switzerland
- Turkey (Türkiye) (2):
  - University Children's Hospital, Adana
  - Cerrahpasa School of Medicine, Istanbul

REFERENCES:
- [Derived] Levai E, Marinovic I, Bartosova M, Zhang C, Schaefer B, Jenei H, Du Z, Drozdz D, Klaus G, Arbeiter K, Romero P, Schwenger V, Schwab C, Szabo AJ, Zarogiannis SG, Schmitt CP. Human peritoneal tight junction, transporter and channel expression in health and kidney failure, and associated solute transport. Sci Rep. 2023 Oct 13;13(1):17429. doi: 10.1038/s41598-023-44466-z. PMID 37833387
- [Derived] Catar RA, Bartosova M, Kawka E, Chen L, Marinovic I, Zhang C, Zhao H, Wu D, Zickler D, Stadnik H, Karczewski M, Kamhieh-Milz J, Jorres A, Moll G, Schmitt CP, Witowski J. Angiogenic Role of Mesothelium-Derived Chemokine CXCL1 During Unfavorable Peritoneal Tissue Remodeling in Patients Receiving Peritoneal Dialysis as Renal Replacement Therapy. Front Immunol. 2022 Feb 4;13:821681. doi: 10.3389/fimmu.2022.821681. eCollection 2022. PMID 35185912
- [Derived] Bartosova M, Zhang C, Schaefer B, Herzog R, Ridinger D, Damgov I, Levai E, Marinovic I, Eckert C, Romero P, Sallay P, Ujszaszi A, Unterwurzacher M, Wagner A, Hildenbrand G, Warady BA, Schaefer F, Zarogiannis SG, Kratochwill K, Schmitt CP. Glucose Derivative Induced Vasculopathy in Children on Chronic Peritoneal Dialysis. Circ Res. 2021 Aug 20;129(5):e102-e118. doi: 10.1161/CIRCRESAHA.121.319310. Epub 2021 Jul 8. PMID 34233458
- See also: International Pediatric Peritoneal Dialysis Network — http://www.pedpd.org